CLINICAL TRIAL: NCT00000779
Title: A Phase I Comparative Blinded Trial of Several HIV-1 Derived Immunogens in Infected Individuals With >= 500 CD4 Cells/mm3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Prevention
Other Study IDs: ACTG 214; 11191 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; Adjuvants, Immunologic; AIDS-Related Complex; HIV Envelope Protein gp120; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Aluminum Hydroxide; MF59 oil emulsion

INTERVENTIONS:
Biological: Aluminum hydroxide
Biological: MF59
Biological: rgp120/HIV-1IIIB
Biological: rgp120/HIV-1MN
Biological: rgp120/HIV-1 SF-2
Biological: Env 2-3

SUMMARY:
PRIMARY: To compare the immunogenicity and safety of each of several HIV-1 derived immunogens versus control in HIV-infected individuals with CD4 counts greater than or equal to 500 cells/mm3.

SECONDARY: To determine whether significant advantages to any one vaccine exist.

Before large clinical trials of anti-HIV vaccines are undertaken, it is important to determine whether there are significant advantages to any one of the vaccines currently offered for such studies.

DETAILED DESCRIPTION:
Before large clinical trials of anti-HIV vaccines are undertaken, it is important to determine whether there are significant advantages to any one of the vaccines currently offered for such studies.

Patients are randomized to receive one of four vaccines or one of two placebo controls. The vaccines are: rgp 120/HIV-1IIIB, rgp 120/HIV-1MN, rgp 120/HIV-1SF, and env 2-3. The two control immunogens are aluminum hydroxide (alum) and BIOCINE Placebo Vaccine 2 (MF-59 adjuvant emulsion in citrate buffer). Patients are vaccinated at weeks 0, 4, 8, 12, 16, 20, 28, and 36. If significant benefit is seen among vaccine patients, then placebo patients may receive vaccination with one of the immunogens producing an immune response.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Short-term nonsteroidal anti-inflammatory therapy.

Patients must have:

* HIV seropositivity.
* CD4 count >= 500 cells/mm3.
* Successful establishment of EBV-transformed B-cell lines at study entry.
* Consent of parent or guardian if < 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Suspected or known allergies to any vaccine components.
* Medical contraindication.
* Problem with compliance.

Concurrent Medication:

Excluded:

* Antiretroviral therapy (e.g., AZT, ddI, or ddC).
* Agents with putative immunomodulating activity (e.g., interferon, steroids, hematopoietin).
* Parenteral therapies (including SC allergy sensitization).
* Other investigational HIV drugs or therapies.

Prior Medication:

Excluded:

* Any prior vaccinations against HIV.
* Antiretroviral therapy (e.g., AZT, ddI, or ddC) within the past 6 months.
* Agents with putative immunomodulating activity (e.g., interferon, steroids, hematopoietin) within the past 3 months.
* Parenteral therapies (including SC allergy sensitization) within the past 3 months.
* Other investigational HIV drugs or therapies within the past 3 months.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Schooley RT, Study Chair; Walker B, Study Chair
Locations (10):
- United States (10):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - NY Univ. HIV/AIDS CRS, New York, New York
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Schooley RT, Spino C, Chiu S, DeGruttola V, Kuritzkes DR. Poor immunogenicity of HIV-1 envelope vaccines with alum or MF59 aduvant in HIV-infected individuals: results of two randomized trials. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:204 (abstract no 756)
- [Background] Schooley RT, Spino C, Kuritzkes D, Walker BD, Valentine FA, Hirsch MS, Cooney E, Friedland G, Kundu S, Merigan TC Jr, McElrath MJ, Collier A, Plaeger S, Mitsuyasu R, Kahn J, Haslett P, Uherova P, deGruttola V, Chiu S, Zhang B, Jones G, Bell D, Ketter N, Twadell T, Chernoff D, Rosandich M. Two double-blinded, randomized, comparative trials of 4 human immunodeficiency virus type 1 (HIV-1) envelope vaccines in HIV-1-infected individuals across a spectrum of disease severity: AIDS Clinical Trials Groups 209 and 214. J Infect Dis. 2000 Nov;182(5):1357-64. doi: 10.1086/315860. Epub 2000 Oct 9. PMID 11023459